CLINICAL TRIAL: NCT03978260
Title: Preoperative Anaemia Prevalence in Surgical Patients- A Prospective, International, Multicentre Observational Study (ALICE)
Brief Title: Preoperative Anaemia prevaLence In surgiCal patiEnts
Acronym: ALICE
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Medical University of Vienna (Other); University Hospital, Angers (Other Government); Medical University of Graz (Other); Hospital del Mar (Other); Hospital Hietzing (Other); University of Zurich (Other); Goethe University (Other); Auckland City Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Patrick Meybohm, M.D., Principal Investigator, Wuerzburg University Hospital
Other Study IDs: E35/19
Record Dates: First submitted 2019-05-23; First posted 2019-06-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Anemia; Iron-deficiency; Folic Acid Deficiency; Vitamin B 12 Deficiency; Anaemia of Renal Disease; Anemia of Chronic Inflammation
Keywords: Anemia
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency; Folic Acid Deficiency; Vitamin B 12 Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Preoperative anaemia is common in surgery, with a prevalence between 10 and 50 %, and is an independent risk factor for morbidity and mortality.

Anaemia is mostly the result of an inadequate erythropoiesis due to iron deficiency, lack of vitamin B12 or folate, and bone marrow diseases. Among the elderly, renal disease and chronic inflammation account for approximately one-third of all anaemia incidences. The aim of this study is to provide detailed data about the prevalence of preoperative deficiencies in iron, vitamin B12 and/or folate and the presence of underlying renal or chronic diseases in patients undergoing major surgery.

DETAILED DESCRIPTION:
Preoperative anaemia is common in surgery, with a prevalence between 10 and 50 %, and is an independent risk factor for morbidity and mortality. Due to the potential risk of additional blood loss, anaemia represents a serious disease condition within the surgical field. Especially patients undergoing major elective surgery are at risk of substantial blood loss. Anaemia is mostly the result of an inadequate erythropoiesis due to iron deficiency, lack of vitamin B12 or folate, and bone marrow diseases. Among the elderly, renal disease and chronic inflammation account for approximately one-third of all anaemia incidences. The aim of this study is to provide detailed data about the prevalence of preoperative deficiencies in iron, vitamin B12 and/or folate and the presence of underlying renal or chronic diseases in patients undergoing major surgery. Results will facilitate design of supplementation strategies to improve haemoglobin level before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent prior to study participating according to the national law requirements
* Patients undergoing major surgery
* Expected hospital stay with a minimum of 24 hours

Exclusion Criteria:

* Preoperative autologous blood donation
* Patients with expected re-surgery within the planned 7-day recruitment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major surgical patients
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of preoperative anaemia | prior surgery
  Hemoglobin level

SECONDARY OUTCOMES:
Number of patients with red blood cell transfusion | 30 day
  Amount of transfused units per patient
Number of patient with revision | 90 day
  Number of patients with Revision after surgery
Number of patients with mortality | 90 day
  in-hospital
Re-admission | up to 90 days after discharge
  Re-admission rates up to 90 days
Hospital and ICU length of stay | 30 days
  Time from Admission till discharge
Incidence of hospital-acquired anaemia | 30 days
  Hemoglobin level

CONTACTS AND LOCATIONS:
Locations (1):
- Johann Wolfgang Goethe University Hospital, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choorapoikayil S, Baron DM, Spahn DR, Lasocki S, Boryshchuk D, Yeghiazaryan L, Posch M, Bisbe E, Metnitz P, Reichmayr M, Zacharowski K, Meybohm P; German Society of Anaesthesiology and Intensive Care (GSAIC) Trials Group; SFAR research network; Supportive Anaesthesia Trainee-led Audit and Research Network (SATURN); ALICE study collaborators. The aetiology and prevalence of preoperative anaemia in patients undergoing major surgery (ALICE): an international, prospective, observational cohort study. Lancet Glob Health. 2025 Dec;13(12):e2041-e2050. doi: 10.1016/S2214-109X(25)00320-1. PMID 41240945